CLINICAL TRIAL: NCT05465915
Title: The Effect of 0.15ms Pulse Width on the Outcome of Electroconvulsive Therapy
Brief Title: Pulse Width 0.15ms vs 0.30ms in Electroconvulsive Therapy
Acronym: PWECT015
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jozef Buday, Head of Neurostimulation Center, General University Hospital in Prague, Charles University, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1885/20 S-IV
Record Dates: First submitted 2022-01-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Major Depressive Disorder; Bipolar Depression
Keywords: Electroconvulsive Therapy, Depression, Pulse-Width
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Subjects are randomized into two groups (blue and red) where crossover titration of ECT is used. From the 3. application and onwards, subjects continue either with 0.15ms or 0.30ms pulse width.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blocked randomization is used to divide patients into blue and red group via an allocator. ECT practitioners are aware which patient belongs to which group but are blinded to block size. Testers, patients and attending psychiatrists are blinded to what group the patients belong to and what ECT parameters are used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Blue (Active Comparator): 1. Session - Titration with 0.30ms pulse width
  2. Session - Titration with 0.15ms pulse width
  3. Session and further - continue with 0.15ms pulse width
  Interventions: Device: Electroconvulsive therapy
- Red (Active Comparator): 1. Session - Titration with 0.15ms pulse width
  2. Session - Titration with 0.3ms pulse width
  3. Session and further - continue with 0.3ms pulse width
  Interventions: Device: Electroconvulsive therapy

INTERVENTIONS:
Device: Electroconvulsive therapy — Patients are treated with ECT.

SUMMARY:
The PWECT015 study was designed to compare the application of 0.15ms and 0.30ms pulse width in electroconvulsive therapy (ECT). Subjects will be compared both within groups and in-group via psychometric scales.

DETAILED DESCRIPTION:
This study is a controlled randomized clinical trial. Patients (projected n=40 are randomized into two groups - blue (20) and red (20). Randomization will be blocked (size sample 4) - 1 allocator. ECT practitioners are aware which patient belongs to which group but are blinded to block size. Testers are blinded to what group the patients belong to and what ECT parameters are used. Patients and attending psychiatrists are also blinded as to which group the patient belongs to.

The MECTA SIGMA device will be used for ECT.

Cross-over titration by stimulation will be used during the application of ECT to find the seizure threshold (ST) as follows:

RED GROUP

1. Session - Titration with 0.15ms
2. Session - Titration with 0.3 ms
3. Session and further - continue with 0.3 ms pulse width and 6x ST found during the second session.

BLUE GROUP

1. Session - Titration with 0.30ms
2. Session - Titration with 0.15ms
3. Session and further - continue with 0.15ms pulse width and 6x ST found during the second session.

Delivered energy is measured in percentage (%) of the maximum charge (in millicoulombs, mC) that the European version of the MECTA SIGMA device is able to administer. Total amount of ECT applications is individual and based on the clinical state of the patient. ECT outcome will be predicted via seizure duration (SD). If the seizure duration is less than 15s, the ECT dosage will be increased during next session by 100%. Throughout the ECT course, patients will be closely monitored by the testers via psychometric scales.

Primary outcome of the study is measured via Time To Recovery (TTR) - which is measured after each ECT application. TTR is the time (in minutes) after which the patient is fully vigilant and aware of his surroundings after an ECT procedure. TTR will be compared both in-group and between groups. Other psychometric measures are specified in the outcome measures section.

ELIGIBILITY:
Inclusion Criteria:

* age equal to 18 or higher
* score equal or higher than 20 on the Montgomery-Asberg Depression Scale (MADRS),
* major depressive disorder or bipolar depression

Exclusion Criteria:

* other axis 1 disorder
* ECT in the last 3 months
* neurological disease
* psychosis
* pregnancy
* any somatic condition that contraindicates ECT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-07-18 (Estimated); Study Completion 2024-01-18 (Estimated)

PRIMARY OUTCOMES:
Time to Recovery (TTR) | immediately after each ECT procedure, measured in minutes.
  time to when the patient is fully vigilant and aware of his surroundings after an ECT procedure
ECCA (Electroconvulsive cognitive assesment) | T1: baseline, 2 days before the commencement of an ECT course, T2: during the course of ECT, between second and third ECT application, T3: after the course of ECT, within 2 days
  cognitive screening optimized for measuring cognitive functions in patients before, during and after the course of ECT.
AMI (Autobiographical Memory Interview) | T1: baseline, 2 days before the commencement of an ECT course, T2: after the course of ECT, within 2 days , T3: 2 months after the ECT course , T4: 4 months after the ECT course, T5: 6 months after the ECT course
  This interview is intended to quantify retrograde amnesia following electroconvulsive therapy (ECT).
MoCA (Montreal Cognitive Assessment) | T1: baseline, 2 days before the commencement of an ECT course, T2: 2 months after the ECT course, T3: 4 months after the ECT course, T4: 6 months after the ECT course
  Screening of cognitive functions, results used as an inclusion criteria of the study and for the determination of the cognitive baseline.
QIDS (The Quick Inventory of Depressive Symptomatology) | T1: baseline, 2 days before the commencement of an ECT course, T2: during the course of ECT, between second and third ECT application, T3: after the course of ECT, within 2 days, T4: 2 months after ECT , T5: 4 months after ECT, T6: 6 months after ECT
  Rates depression symptoms via self-assessment
MADRS (Montgomery-Asberg Depression Rating Scale) | T1: baseline, 2 days before the commencement of an ECT course, T2: during the course of ECT, between second and third ECT application, T3: after the course of ECT, within 2 days, T4: 2 months after ECT , T5: 4 months after ECT, T6: 6 months after ECT
  Assessment of depression severity, objective scale based on clinicians interview with a patient, results also used as an inclusion criteria of the study.
BVMT-R (Brief Visuospatial Memory Test-Revised) | 1: baseline, 2 days before the commencement of an ECT course, T2: after the course of ECT, within 2 days , T3: 2 months after the ECT course , T4: 4 months after the ECT course, T5: 6 months after the ECT course
  Neuropsychological assessment designed to evaluate visuospatial memory in patients.
RAVLT (The Rey Auditory Verbal Learning Test) | 1: baseline, 2 days before the commencement of an ECT course, T2: after the course of ECT, within 2 days , T3: 2 months after the ECT course , T4: 4 months after the ECT course, T5: 6 months after the ECT course
  Neuropsychological assessment designed to evaluate verbal memory in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Heidingerová, Principal Investigator — Department of Psychiatry, First Faculty of Medicine, Charles University
Locations (1):
- Psychiatric Department, General University Hospital and 1st Faculty of Medicine, Prague, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon request from a verified researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after the end of study, indefinitely
Access Criteria: upon individual request by a verified researcher